CLINICAL TRIAL: NCT02294565
Title: A Phase I/II Study of VST-1001 (Dilute Fluorescein) for Lymphatic Mapping and Localization of Lymph Nodes Draining a Primary Tumor Site in Patients With Clinically Node Negative Breast Cancer
Brief Title: VST-1001 (Dilute Fluorescein) for Lymphatic Mapping & Localization of Lymph Nodes in Patients With Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vestan, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other); Huntsman Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: VST-1001-02; 2013-1021 (Other: The University of Texas M.D. Anderson Cancer Center)
Record Dates: First submitted 2014-10-22; First posted 2014-11-19 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Breast Cancer
Keywords: Sentinel Lymph Node Biopsy; Breast Cancer; Lymphatic Mapping
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VST-1001 & 99mTc-labeled sulfur colloid (Other): VST-1001 (with medical devices) and 99mTc-labeled sulfur colloid are used together during a SLNB procedure in a single subject. Both drugs are evaluated for lymphatic mapping and localization of lymph nodes. The current standard of care for lymphatic mapping and lymph node localization during a SLNB procedure is a combined-modality technique that employs both a radiotracer (99mTc-labeled sulfur colloid is the radiotracer used in this study) and a vital blue dye (a patient receives both drugs). In this study, the vital blue dye is replaced with VST-1001 and companion medical devices.
  VST-1001 is excited by a medical device (blue-light LED illuminator) to fluoresce; the surgeon is wearing blue-light filtering eyewear to improve visualization of the relevant tissue structures.
  Interventions: Drug: VST-1001; Drug: 99mTc-labeled sulfur colloid

INTERVENTIONS:
Drug: VST-1001 — Single-dose injection (peritumoral, periareolar, and/or intradermal) of VST-1001 administered pre-SLNB procedure; VST-1001 is used with medical devices (blue-light LED illuminator and blue-light filtering eyewear) for lymphatic mapping and localization of lymph nodes during a SLNB procedure.
  Other Names: dilute fluorescein
Drug: 99mTc-labeled sulfur colloid — Single-dose injection (peritumoral, periareolar, intradermal, and/or subdermal) of 99mTc-labeled sulfur colloid administered per standard of care; the radioactivity of the radioactive colloid is detected with a gamma probe per standard of care.
  Other Names: radiocolloid; radiotracer

SUMMARY:
The purpose of this Phase 1 portion of this clinical research study is to find out what dose of dilute fluorescein is needed for a surgeon to best see important lymph nodes that need to be removed during surgery (a standard of care surgery referred to as a Sentinel Lymph Node Biopsy procedure) in patients diagnosed with breast cancer.

The purpose of the Phase 2 portion of this clinical research study is to find out if giving dilute fluorescein sodium in combination with a radiotracer (a drug that is radioactive) can help surgeons localize the lymph nodes that need to be removed in patients diagnosed by breast cancer.

DETAILED DESCRIPTION:
The study is a single center prospective, non randomized, single arm, open label, single dose VST-1001 study for lymphatic mapping and localization of lymph nodes draining a primary tumor site in patients with clinically node negative breast cancer.

This study evaluates the combined modality technique of investigational VST-1001 with companion medical devices (replacing the blue dye) and 99mTc-labeled sulfur colloid for concordance in lymphatic mapping and localization of lymph nodes in patients who are undergoing a sentinel lymph node biopsy (SLNB) surgical procedure.

This purpose of the Phase I study is to determine a safe and effective recommended dose of VST-1001 for intraoperative lymphatic mapping and localization of lymph nodes draining a breast tumor. The purpose of the Phase II study is to further evaluate the Phase I study recommended dose of VST-1001 and to evaluate its ability to provide intraoperative visualization of the lymphatic system and lymph nodes draining the primary tumor in patients diagnosed with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary breast cancer.
* Diagnosed with invasive adenocarcinoma, or DCIS for which a SLNB is the recommended standard of care, or breast cancer with all of the following conditions met:

  * FNA results positive for cancer cells
  * positive clinical breast examination
  * mammography and/or US and/or MRI abnormality(ies) consistent with malignancy.
* N0 and M0 at the time of study entry.
* ECOG 0, 1, or 2

Exclusion Criteria:

* A tumor with direct extension to the chest wall and/or to the skin.
* Diffuse tumors or multiple malignant tumors in the breast.
* Prior breast malignancy of the ipsilateral breast.
* Patient currently receiving or had prior treatment for the currently diagnosed breast cancer.
* Medical conditions and/or prior surgical procedures that have the potential to substantially alter the lymphatic drainage pattern from the primary tumor to the lymph node basin.
* Inability to localize 1 or 2 lymph node drainage basin(s) via lymphatic mapping.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
LYMPH NODE-LEVEL CONCORDANCE of Visually Observed VST-1001 Fluorescence and 99mTc-Labeled Sulfur Colloid Radioactivity, where CONCORDANCE is defined relative to radioactive nodes | The primary outcome is assessed during surgery.
  Fluorescence and radioactivity data will be collected during the SLNB surgical procedure.

SECONDARY OUTCOMES:
LYMPH NODE-LEVEL REVERSE CONCORDANCE of Visually Observed VST-1001 Fluorescence and 99mTc-Labeled Sulfur Colloid Radioactivity, where REVERSE CONCORDANCE is defined relative to fluorescent nodes | The secondary outcome is assessed during surgery.
  Fluorescence and radioactivity data will be collected during the SLNB surgical procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Robert HI Andtbacka, MD, Study Director — Vestan, Inc.; Merrick I Ross, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas
  - The University of Utah Huntsman Cancer Institute, Salt Lake City, Utah